CLINICAL TRIAL: NCT00961129
Title: The Continuing Care Needs From Receiving Treatment to Survival in Colorectal Cancer Patients in Different Stages
Brief Title: The Continuing Care Needs in Colorectal Cancer Patients in Different Stages
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Shiow-Ching Shun, Assistant Professor, National Taiwan University
Other Study IDs: 200902016R
Record Dates: First submitted 2009-08-16; First posted 2009-08-18 (Estimated); Last update posted 2010-04-13 (Estimated); Status verified 2010-04

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer; needs; survivors; any stage
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- patients with colorectal cancer: patients with colorectal cancer in any stage or survivors

SUMMARY:
The aims of this study are to:

1. explore supportive care needs in colorectal cancer patients with treatment and survivors;
2. compare the supportive care needs in different stage of colorectal cancer;
3. identify the significant factors for the supportive care needs;
4. explore the supportive care needs within one year after newly diagnosis.

DETAILED DESCRIPTION:
Both large scale cross-sectional survey and a prospective 1-year longitudinal panel study design will be used in this study. The cross-sectional survey is to examine the current status of supportive care needs perceived by different stage of colorectal cancer inpatients and outpatients including survivors. The 1-year longitudinal design is to explore the change of supportive care needs perceived by patients within one year after newly diagnosed with colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients with colorectal cancer in any stage or survivors
* Those who are willing to participate in the research
* Aged above 18

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: recruit colon cancer inpatients and outpatients in clinics
Sampling Method: Non-Probability Sample
Enrollment: 269 (Estimated)
Dates: Start 2009-03; Primary Completion 2010-04 (Actual); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
supportive cancer care needs | For 1-year follow-up study, measurement time-points include 1, 3, 6, 9, and 12 months after diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: shiow-ching shun, PhD, Principal Investigator — National Taiwan University
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan